CLINICAL TRIAL: NCT03238209
Title: Correlation and Compatibility Between Surface Respiratory Electromyography and Transesophageal Diaphragmatic Electromyography Measurements During Treadmill Exercise in Stable Patients With COPD
Brief Title: Surface Respiratory Electromyography Measurements During Treadmill Exercise in Stable Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weiliang Wu, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GuangzhouInsReD
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Respiratory Disease
Keywords: neural respiratory drive; transesophageal diaphragmatic EMG; surface diaphragmatic EMG; surface sternocleidomastoid EMG; surface parasternal intercostal muscle EMG
MeSH Terms: conditions — Respiration Disorders | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise testing (Experimental): The test consisted of a steady-state resting period of 3 min followed by 1 min of unloaded pedaling at 60 cycles/min for each individual; the exercise load was increased by 10 W each min until the test had to be stopped because symptoms prevented further exercise. After test results were recorded, EMGdi,es and each surface inspiratory EMG of maximal exercise capacity were analysed.
  Interventions: Diagnostic Test: Exercise testing

INTERVENTIONS:
Diagnostic Test: Exercise testing — The test consisted of a steady-state resting period of 3 min followed by 1 min of unloaded pedaling at 60 cycles/min for each individual; the exercise load was increased by 10 W each min until the test had to be stopped because symptoms prevented further exercise. After test results were recorded, EMGdi,es and each surface inspiratory EMG of maximal exercise capacity were analysed.

SUMMARY:
To evaluate the compatibility and correlation between noninvasive surface respiratory electromyography and invasive transesophageal diaphragmatic electromyography measurements, as facilitating indicators of neural respiratory drive evaluation during treadmill exercise. Transesophageal diaphragmatic EMG (EMGdi,es) and surface inspiratory EMG, including surface diaphragmatic EMG (EMGdi,sur), surface parasternal intercostal muscle EMG (EMGpara) and surface sternocleidomastoid EMG (EMGsc) were detected simultaneously during increasing capacity exercise in stable patients with COPD. EMGdi,es, EMGdi,sur, EMGpara and EMGsc was quantified using root mean square (RMS), which represent as RMSdi,es, RMSdi,sur, RMSpara and RMSsc.

DETAILED DESCRIPTION:
Subjects This self-matching clinical trial included twenty patients with COPD (age range, 40-80 years) treated at outpatient respiratory medicine departments at the First Affiliated Hospital of Guangzhou Medical University between July 2016 and December 2016. The diagnosis of COPD in all participants were measured using the pulmonary spirometry, according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD).1 Inclusion criteria: 1) post bronchodilator forced expiratory volume in 1 s [FEV1]/forced vital capacity [FVC] ,70% and FEV1 ,50% of the predicted value); 2) bronchial dilation test (BDT) negative. Exclusion criteria: 1) acute exacerbation in the previous 4 weeks; 2) use of oral corticosteroids within 4 weeks; and 3) smoking more than 10 cigarettes daily; (4) history of other respiratory, cardiovascular, neuromuscular, and musculoskeletal diseases that could interfere with the exercise performance and inspiratory muscle activities.

Study design This study has been reviewed and published on the ClinicalTrials.gov public site (identifier: NCT03017300, Clinical trial date of registration: March 29, 2017). The study protocol was approved by the Ethics Committee of the First Affiliated Hospital of Guangzhou Medical University. Informed consent was obtained from COPD patients before participation in this study. To ensure the rights of all participants were protected, the researchers strictly adhered to the Declaration of Helsinki and the ethical principles in designing and conducting clinical research.

Measurements of transesophageal diaphragmatic EMG (EMGdi,es) EMGdi,es is the classic representative index describing activity of diaphragmatic myoelectric signals, the electrical manifestations of the excitation process elicited by action potentials propagating along muscle fiber membranes. The EMG signal is detected with multiple electrodes and then amplified, filtered, and displayed on a screen or digitized to facilitate further analysis. Electromyography of respiratory muscles can be used to assess the level and pattern of their activation so as to detect and diagnose neuromuscular pathology and, when coupled with tests of mechanical function, to assess the efficacy of the muscle's contractile function. Neural respiratory drive, expressed as EMGdi, was measured using a multipair esophageal electrode consisting of nine consecutive coils composed of five electrode pairs positioned in the esophagus and traversing the cardia. EMGdi signals acquired with digital sampling at 2 kHz were bandpass filtered (10 Hz-3 kHz) and amplified. Peak RMS per respiratory cycle was calculated and averaged over 1 min. RMS of the EMGdi signal is thequantification of the total EMGdi power. Theoretically, the RMS of the EMGdi reflects the force output from the brainstem respiratory centre to the peripheral respiratory muscles and also reflect the sensation of dyspnea.

Measurements of surface inspiratory EMG EMG electrodes The electrical activity of the surface inspiratory EMG was derived transcutaneously from pairs of single disposable electrodes (Neotrode, Conmed Corporation, New York, USA). For the commonor ground electrode the same disposable electrode was used. Electrical activity of the sternocleidomastoidmuscles and Intercostals muscles were derived transcutaneously from reusablebipolar electrodes formed by two narrow rim electrodes housings, each containing a 4mm Ag-AgCl sintered electrode pallet (InVivo Metrics, Healdsburg, USA), interconnected with a plastic clip (homemade UMCG, Groningen, The Netherlands) at a distance of14mm. After filling the electrode cavity with electrode gelthe assembly was fixed to the skin by means of double sided adhesives. All EMG signals detected by electrodes were convey to connected to the biological signal acquisition and analysis system (Powerlab 16/35; ADInstruments) by shielded low noise cables.

Electrode placement Surface diaphragmatic EMG (EMGdi,sur): The surface detecting electrode couple were separately placed at the intersection point of the sixth and eight intercostal space and anterior axillary line, at a distance of 5 cm.10 Surface parasternal EMG (EMGpara): The surface detecting electrodes were placed bilaterally in the second intercostal space, about 3 cm parasternal, a reference ground electrode was placed atthe sternum sternal angle.

Surface sternocleidomastoid EMG (EMGsc): Surface detecting electrode were placed on the 1/3 and 2/3 of overall length of sternocleidomastoid, a reference ground electrode was placed at the suprasternal fossa.

Exercise testing All subjects performed a maximal incremental cycle ergometry test in a sitting posture, in order to minimize the effects of muscle activity necessary for body stabilization (Ergoselect 200 K; Cosmed, Rome, Italy). Furthermore, to minimize muscle activity for head positioning, the subjects were instructed to look straight ahead during the measurements. The test consisted of a steady-state resting period of 3 min followed by 1 min of unloaded pedaling at 60 cycles/min for each individual; the exercise load was increased by 10 W each min until the test had to be stopped because symptoms prevented further exercise. After test results were recorded, EMGdi,es and each surface inspiratory EMG of maximal exercise capacity were analysed.

ELIGIBILITY:
Inclusion criteria:

1. post bronchodilator forced expiratory volume in 1 s [FEV1]/forced vital capacity [FVC] ,70% and FEV1 ,50% of the predicted value);
2. bronchial dilation test (BDT) negative.

Exclusion criteria:

1. acute exacerbation in the previous 4 weeks;
2. use of oral corticosteroids within 4 weeks;
3. smoking more than 10 cigarettes daily;
4. history of other respiratory, cardiovascular, neuromuscular, and musculoskeletal diseases that could interfere with the exercise performance and inspiratory muscle activities.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
transesophageal diaphragmatic EMG | 30 minute
  transesophageal diaphragmatic EMG was measured using a multipair esophageal electrode consisting of nine consecutive coils composed of five electrode pairs positioned in the esophagus and traversing the cardia

SECONDARY OUTCOMES:
Surface diaphragmatic EMG | 30 minute
  The surface detecting electrode couple were separately placed at the intersection point of the sixth and eight intercostal space and anterior axillary line, at a distance of 5 cm.
Surface parasternal EMG | 30 minute
  The surface detecting electrodes were placed bilaterally in the second intercostal space, about 3 cm parasternal, a reference ground electrode was placed atthe sternum sternal angle.
Surface sternocleidomastoid EMG | 30 minute
  Surface detecting electrode were placed on the 1/3 and 2/3 of overall length of sternocleidomastoid, a reference ground electrode was placed at the suprasternal fossa.